CLINICAL TRIAL: NCT06660576
Title: Histochemical Analysis of Gallbladder Stones in Children and Correlation With Etiological Factors
Brief Title: Gallbladder Stones in Children and Correlation With Etiological Factors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hitham Diaaeldin Ahmed, M.B.B.Ch., Resident of Pediatric Surgery Sohag University Hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-15-10-7MS
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Gallbladder Stone
MeSH Terms: conditions — Cholecystolithiasis | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gallbladder stones in children (Other): Histochemical analysis of Gallbladder stones in children and correction with aetiological factors
  Interventions: Procedure: Cholecystectomy and histochemical analysis of Gallbladder stones

INTERVENTIONS:
Procedure: Cholecystectomy and histochemical analysis of Gallbladder stones — Cholecystectomy and histochemical analysis of Gallbladder stones

SUMMARY:
Aims of the Study:

The objective of this study is to estimate the correlation between etiological factors and postoperative histochemical analysis of pediatric gallbladder stones.

DETAILED DESCRIPTION:
Study design:

A prospective, cohort study. Duration of the study: The study starts from October 2024 to August 2025.

Place of the study:

The study will be held in Department of Pediatric surgery in Sohag University Hospital.

Inclusion and exclusion criteria:

Inclusion criteria:

Age <18 years . Symptomatic gallbladder stones (biliary colic, fever, vomiting, positive Murphy sign ) .

Congenital hemolytic anemia with gallbladder stones. Asymptomatic patient with gallbladder stones <5mm after medical treatment (Ursodeoxycholic acid ) for 1year .

Imaging criteria ( large gallbladder stone < 1cm diameter , gallbladder thickness >3mm ) either symptomatic or asymptomatic .

Exclusion criteria:

Age >18 years. Asymptomatic patients who improved after follow up and medical treatment . Biliary anomaly as choledochal cyst , biliary stricture. Common bile duct stones .

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

Age <18 years . Symptomatic gallbladder stones (biliary colic, fever, vomiting, positive Murphy sign ) .

Congenital hemolytic anemia with gallbladder stones. Asymptomatic patient with gallbladder stones <5mm after medical treatment (Ursodeoxycholic acid ) for 1year .

Imaging criteria ( large gallbladder stone < 1cm diameter , gallbladder thickness >3mm ) either symptomatic or asymptomatic .

Exclusion Criteria:

* Age >18 years. Asymptomatic patients who improved after follow up and medical treatment . Biliary anomaly as choledochal cyst , biliary stricture. Common bile duct stones .

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Early follow up to detect aetiology of gallbladder stones | One week after operation
  Aetiology of gallbladder stones

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Background] Buch S, Schafmayer C, Volzke H, Becker C, Franke A, von Eller-Eberstein H, Kluck C, Bassmann I, Brosch M, Lammert F, Miquel JF, Nervi F, Wittig M, Rosskopf D, Timm B, Holl C, Seeger M, ElSharawy A, Lu T, Egberts J, Fandrich F, Folsch UR, Krawczak M, Schreiber S, Nurnberg P, Tepel J, Hampe J. A genome-wide association scan identifies the hepatic cholesterol transporter ABCG8 as a susceptibility factor for human gallstone disease. Nat Genet. 2007 Aug;39(8):995-9. doi: 10.1038/ng2101. Epub 2007 Jul 15. PMID 17632509
- [Background] Wesdorp I, Bosman D, de Graaff A, Aronson D, van der Blij F, Taminiau J. Clinical presentations and predisposing factors of cholelithiasis and sludge in children. J Pediatr Gastroenterol Nutr. 2000 Oct;31(4):411-7. doi: 10.1097/00005176-200010000-00015. PMID 11045839
- [Background] Curro G, Meo A, Ippolito D, Pusiol A, Cucinotta E. Asymptomatic cholelithiasis in children with sickle cell disease: early or delayed cholecystectomy? Ann Surg. 2007 Jan;245(1):126-9. doi: 10.1097/01.sla.0000242716.66878.23. PMID 17197975